CLINICAL TRIAL: NCT00139828
Title: Post Marketing Study in Haemophilia B Patients Using Nonafact® 100 IU/ml Powder and Solvent for Solution for Injection(Human Coagulation Factor IX)(Human Plasma Derived Factor IX Product, Freeze Dried)
Brief Title: Post Marketing Study in Haemophilia B Patients Using Nonafact® (Human Coagulation Factor IX)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB2000.03
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: Hemophilia B
Keywords: haemophilia B; factor IX; Product Surveillance, Postmarketing; plasma products
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): The amount of Nonafact® to be administered and the frequency of treatment is based on the SmPC and should always be determined on the basis of the clinical effectiveness in the individual patient
  Interventions: Drug: human coagulation Factor IX

INTERVENTIONS:
Drug: human coagulation Factor IX
  Other Names: Nonafact

SUMMARY:
In this postmarketing study, the safety of Nonafact® (human coagulation factor IX) is evaluated in previous treated and untreated patients with severe, moderate or mild haemophilia B.

DETAILED DESCRIPTION:
The clinical efficacy and safety of Nonafact® has been shown in two pre-authorisation studies. Marketing authorisation for the EU was granted 3 July 2001. The Post Marketing Study, which evaluates the clinical efficacy, immunogenicity and safety of Nonafact®, is set up according to CPMP/BPWG /198/95, rev. 1 (Final, London, 19 October 2000) 'Note for guidance on the clinical investigation of human plasma derived factor VIII and IX products'

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia B (mild, moderate or severe), Haemophilia B Leyden or symptomatic carriers of Haemophilia B and Haemophilia B Leyden
* Above the age of six, at the moment of inclusion
* Tested positive for HAV and HBV antibodies, induced by infection or vaccination, and negative for HBsAg
* Informed consent signed by the patients or his legally accepted representative

Exclusion Criteria:

* Under the age of six, at the moment of inclusion
* Tested negative for HAV and HBV antibodies

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Number of bleeding episodes (efficacy after administration) | 24 months
Haematological variables and clinical chemistry (safety) | 24 months
Adverse events (safety) | 24 months

SECONDARY OUTCOMES:
Occurrence of antibodies to factor IX | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: E P Mauser-Bunschoten, MD, PdD, Principal Investigator — UMC Utrecht, Van Creveldkliniek, Utrecht, The Netherlands
Locations (7):
- Netherlands (7):
  - Academic Medical Centre, Amsterdam
  - Kennemer Gasthuis, Haarlem
  - LUMC, Leiden
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Centre, Rotterdam
  - Leyenburg Hospital, The Hague
  - Van Creveldkliniek, Utrecht